CLINICAL TRIAL: NCT04813471
Title: Managing Endothelial Dysfunction in Critically Ill COVID-19 Patients at the Lebanese American University Medical Center- Rizk Hospital
Brief Title: Managing Endothelial Dysfunction in Critically Ill COVID-19 Patients at LAUMCRH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese American University Medical Center (Other)
Responsible Party: Principal Investigator, Kamal Matli, Cardiology Fellow, Lebanese American University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAUMCRH
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Endothelial Dysfunction
MeSH Terms: conditions — COVID-19 | interventions — Nicorandil; Atorvastatin; Folic Acid; Vitamin B Complex

STUDY DESIGN:
Intervention Model Description: Open label Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endothelial Dysfunction Protocol (Experimental): Experimental: Endothelial Dysfunction Protocol
  Our study will evaluate the impact of the endothelial treatment protocol (atorvastatin(or home statin), nicorandil, l-arginine, folic acid and vitamin B complex) in critically Ill patients already on optimal medical therapy for the treatment of COVID-19 virus. Protocol will be given for a total of 14 days or until discharge from the hospital
  Patients already on home statin will continue their medication or if the are eligible for statins they will recieve 40 mg tablet to be given PO once daily.
  Nicorandil Nicorandil 10 mg PO BID for the first 7 days and then if no contraindications escalated to 20 mg PO BID for the remaining 7 days
  Folic Acid Folic Acid 5 mg po once daily
  L-Arginine L-Arginine 1 g po TID
  Vitamin B complex (Becozyme) 1 ampoule IV daily
  Interventions: Drug: Endothelial Protocol
- Standard of care (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Endothelial Protocol — Endothelial Protocol
  Other Names: nicorandil; Atorvastatin or home statin; Folic acid; vitamin B complex; L-argining
  Arms: Endothelial Dysfunction Protocol

SUMMARY:
COVID-19 Infection has been found to cause endothelial dysfunction and most of the adverse events stem to this mechanism. So we seek to target endothelial dysfunction in critically Ill patients with covid by giving them an endothelial protocol ( L-arginine, Folic Acid, Statin, Nicorandil, Vitamin B complex) and monitor clinical outcome in those patients.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) is the novel pathogen responsible for coronavirus disease 2019 (COVID-19) first discovered in Wuhan, China [1]. Since its emergence in late December 2019, many pathophysiological mechanisms have been proposed with multiple pathways that involve various organ systems [2, 3]. Although considered at its emergence as a respiratory infection with manifestations ranging from lower respiratory tract infection to pneumonia and advancing to acute respiratory disease syndrome (ARDS) in its final stages, recent evidence has highlighted how disseminated the virus can be affecting almost every organ be it the heart, kidneys, or blood vessels . Recent trends in research have focused on elucidating the cardiovascular dysfunction in COVID-19 patients especially following studies showing that cardiovascular risk factors are among the most common presenting comorbidities and that cardiovascular complications of SARS-CoV-2 are among the most lethal [4-11] . Initial research revealed that the virus makes use of the angiotensin-converting enzyme 2 (ACE-2) receptor, a widely expressed receptor found in multiple cells lining the lung, heart, gastrointestinal tract, kidneys and endothelial cells to infiltrate host cells. Another prominent mechanism of infection is immune system dysregulation manifesting as a cytokine storm and inflammatory response over-activation [12, 13].

Attempts at laying out a comprehensive or unifying pathogenesis of a COVID-19 infection have singled out endothelial dysfunction as a core pathway [14]. The endothelium is a monolayer of squamous endothelial cells lining the inner surface of arteries, veins and microvasculature. The endothelium hence plays a major role in homeostasis with interactive roles in blood pressure regulation, anti-coagulation and immune protection. Moreover, it is relevant to note that the most common comorbidities that present with COVID-19 such as hypertension, diabetes, obesity and old age are all underlined by pre-existing endothelial damage or dysfunction. As such, endothelial dysfunction and oxidative stress and their relation to the manifestation and progression of COVID-19 infections has gained significant traction in recent publications [15]. This breakthrough exposes several causes of endothelial dysfunction which include direct lining attack, hypoxia, cytokine storm and suppressed endothelial nitric oxide synthase (eNOS) with concomitant nitric oxide deficiency [15]. Several studies have emphasized the role of Nitric Oxide (NO) signaling as a major regulator of vascular tone with its antioxidant, anti-inflammatory and antithrombotic activity. For example, augmenting the production of NO and its bioavailability by Nicorandil has been proposed as a potential treatment in patients with COVID 19. Nicorandil is a vasodilatory agent composed of N-[2-hydroxyethyl]-Nicotinamide Nitrate) used among patients with acute heart failure emergencies. However, it has never been tested in patients with cardiovascular complications resulting from COVID 19 [16]. Moreover, statins are cardio-protective in nature with recent reports showing that they can be beneficial in COVID-19 [17]. An important mechanism via which Statins may improve endothelial function include increasing the production of NO and subsequent vasodilation effect, along with its established major anti-inflammatory and anti-oxidant properties [17]. Vitamin B complex will be used because of the role it plays in cell functioning, energy metabolism, and proper immune function. In addition of its assistance in proper activation of the immune response, reducing pro-inflammatory cytokine levels, improving respiratory function, maintaining endothelial integrity, preventing hypercoagulability and reducing the length of stay in hospital. [18-19-20] Furthermore, eNOS overexpression leads to an increase in NO formation only when the BH4 synthase GTP-cyclohydrolase 1 (GCH-1) is also up-regulated. So, Folic Acid and L-arginine will be given to supplement our patients with BH4 (Tetrahydrobiopterin) [21]. We hypothesize that its administration along with the other previously mentioned agents would improve endothelial function in patients suffering from COVID 19 via a cumulative increase in the bioavailability of NO, and thus improving patients' outcomes

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must have a PCR confirming COVID 19 status
* Participants must be classified as critical as per the FDA evidence of critical illness, which is defined as respiratory failure requiring at least one of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high- flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)
* Eligible for or already taking Statin

Exclusion Criteria:

* Patients who are already on statins or Nicorandil.
* Patients labeled as having mild, moderate or severe COVID-19 infection as per the FDA definitions.
* Patients with shock as defined by SBP<90 for more than 30 minutes not responding to IV fluids with evidence of end organ damage.
* Severe hepatic impairment (Child-Pugh class C) or active liver disease are absolute reasons not to be included especially those with unexplained persistent elevations of serum transaminases.
* Pregnancy or breastfeeding
* Hypersensitivity to any of the above-mentioned medications
* On Levodopa.
* Patients on PDE5 inhibitors, Riociguat
* Acute pulmonary edema
* Hypovolemia
* Leber's disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | will followed up for a total of 28 days
  Clinical improvement was defined as improvement of at least two points from the baseline from date of intervention administration until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 1-month status on the six-category ordinal scale. This scale contains the subsequent categories: (1) death (2) hospital admission requiring invasive mechanical ventilation (3) hospital admission, requiring non-invasive positive pressure ventilation (4) hospital admission, requiring oxygen (5) hospital admission, not requiring oxygen (6) discharge

SECONDARY OUTCOMES:
Need for invasive mechanical ventilation | F/up for 28 days
Length of ICU stay | F/up for 28 days
Length of hospital Stay | F/up for 28 days
Length of need of mechanical ventilation | F/up for 28 days
All cause mortality | F/up for 28 days
Occurrence of side effects | F/up for 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- LAUMCRH, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No